CLINICAL TRIAL: NCT01053546
Title: Effects of Early vs Late Onset of Swallowing Exercises on Patients Undergoing Radiation Treatment for Head and Neck Cancer
Brief Title: Effects of Swallowing Exercises on Patients Undergoing Radiation Treatment for Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00010437; NCI-2009-01445 (Other: CTRP); CCCWFU 98109 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer; Stage I Hypopharyngeal Cancer; Stage I Laryngeal Cancer; Stage I Oropharyngeal Cancer; Stage II Hypopharyngeal Cancer; Stage II Laryngeal Cancer; Stage II Oropharyngeal Cancer; Stage III Hypopharyngeal Cancer; Stage III Laryngeal Cancer; Stage III Oropharyngeal Cancer; Stage IV Hypopharyngeal Cancer; Stage IV Laryngeal Cancer; Stage IV Oropharyngeal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Early exercise group) (Experimental): Patients perform swallowing exercises comprising lingual press, head lift, breath hold, Masako swallow, high pitch e, effortful swallow, and neck stretch and massage for 2 weeks prior to beginning radiotherapy and again immediately after completion of radiotherapy.
  Interventions: Behavioral: exercise intervention; Other: questionnaire administration; Procedure: quality-of-life assessment
- Arm II (Late exercise group) (Experimental): Patients begin performing swallowing exercises as in arm I 1 month after completion of radiotherapy.
  Interventions: Behavioral: exercise intervention; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Behavioral: exercise intervention — The early exercise group will start study exercises approximately two weeks prior to the onset of XRT. The late exercise group will start study exercises one month after the completion of XRT. Participants will undergo an initial/pre-radiation and 1-, 3-, 6-, and 12 month post-radiation swallowing assessments.
Other: questionnaire administration — Ancillary study
Procedure: quality-of-life assessment — Ancillary study
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Swallowing exercise therapy may improve the quality of life of head and neck cancer patients undergoing chemotherapy or radiation therapy.

PURPOSE: This randomized phase III trial is studying early onset of swallowing exercise therapy to see how well it works compared to late onset of swallowing exercise therapy in treating patients with head and neck cancer undergoing chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the difference between early and late onset swallowing exercises on swallowing quality of life in patients undergoing chemo/radiation therapy for head and neck cancer.

SECONDARY OBJECTIVE:

I. To assess the difference between early and late onset swallowing exercises on swallowing function in patients undergoing radiation therapy for head and neck cancer.

TERTIARY OBJECTIVE:

I. To assess the difference between early and late onset swallowing exercises on: individual domains of swallowing quality of life; Penetration Aspiration Scale (PAS) as assessed via FEES; diet level (Dysphagia Outcome and Severity Scale (DOSS) as assessed via FEES; feeding tube duration (days); Eating Assessment Tool (EAT); lingual strength as assessed via lingual manometry; and percent weight loss and percent weight recovery.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I (Early exercise group): Patients perform swallowing exercises comprising lingual press, head lift, breath hold, Masako swallow, high pitch e, effortful swallow, and neck stretch and massage for 2 weeks prior to beginning radiotherapy and again immediately after completion of radiotherapy.

Arm II (Late exercise group): Patients begin performing swallowing exercises as in arm I 1 month after completion of radiotherapy.

In both arms, swallowing exercises are performed twice daily, 6 days a week, for 12 months following completion of radiotherapy.

ELIGIBILITY:
Inclusion

* Written informed consent must be obtained from all participants prior to beginning therapy (participants should have the ability to understand be willing to sign a written informed consent document)
* Individuals with oropharyngeal, hypopharyngeal, or laryngeal cancer of Stages I-IV undergoing radiation and chemo therapies at Wake Forest Baptist Medical Center
* Participants will have surgically received no more than selective neck dissection and tumor biopsy (participants who have undergone primary tumor resection or radical neck dissection will not be eligible)
* Participants must have completed a minimum of third grade education in order to answer questions of the quality of life survey
* Participants must be willing to participate in the swallowing exercise program

Exclusion

* Medical history of cerebrovascular accident, Parkinson's disease, any type of dementia, myasthenia gravis, or amyotrophic lateral sclerosis
* Previous radiation treatment for head/neck cancer
* Swallowing problem of etiology other than current lesion
* Pregnant women are not anticipated in the patient population, but would be excluded from participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
M.D. Anderson Dysphagia Inventory (MDADI) swallowing quality of life score | Baseline and at 1, 3, 6, and 12 months following completion of radiotherapy

SECONDARY OUTCOMES:
Penetration Aspiration Scale (PAS) as assessed via FEES | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Diet level (Dysphagia Outcome and Severity Scale (DOSS)) as assessed via FEES | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Feeding tube duration (days) | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Eating Assessment Tool (EAT) quality of life score | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Lingual strength as assessed by lingual manometry | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Percent weight loss | Baseline and at 1, 3, and 6 months following completion of radiotherapy
Percent weight recovery | Baseline and at 1, 3, and 6 months following completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Susan Butler, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States